CLINICAL TRIAL: NCT02362516
Title: Non-randomised, Open Label, Sequential-group Study to Assess the Pharmacokinetics and Pharmacodynamic Effect of Different Multiple Oral Doses of BI 425809 in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamic Effect of Different Multiple Oral Doses of BI 425809
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346.3; 2014-005652-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

ARMS (1):
- BI 425809 (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809
  Other Names: Iclepertin

SUMMARY:
To assess the exposure of BI 425809 in cerebrospinal fluid relative to plasma as well as safety and tolerability, and to evaluate the effect of different doses of BI 425809 on biomarkers levels in cerebrospinal fluid.

ELIGIBILITY:
Inclusion criteria:

* Healthy male according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), puls rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including blood pressure (BP), puls rate (PR) or electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range and considered as clinical relevant by investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders Further exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUC0-14 (area under the concentration-time curve of the analyte in plasma and CSF over the time interval from 0 to 14h) | 17 days
Cmax (maximum measured concentration of the analyte in plasma and CSF) | 17 days
C312 (concentration of the analyte in plasma and CSF at the time point 312h) | 17 days

SECONDARY OUTCOMES:
frequency [N(%)] of subjects with drug-related adverse events (AEs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.3.32001 Boehringer Ingelheim Investigational Site, Antwerp, Belgium